CLINICAL TRIAL: NCT01608867
Title: A Phase 1 Dose Escalation Study of OMP-54F28 in Subjects With Solid Tumors
Brief Title: A Dose Escalation Study of OMP-54F28 in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54F28-001
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Solid Tumors
Keywords: Phase 1; dose escalation; histologically confirmed; malignancy; metastatic
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — OMP-54F28

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: OMP-54F28 — dose escalation of 0.5, 1, 2.5, 5, and 10 mg/kg administered IV once every 3 weeks

SUMMARY:
This is an open-label Phase 1 dose escalation study of OMP-54F28 in subjects with a solid tumor for which there is no remaining standard curative therapy. Subjects will be assessed for safety, immunogenicity, pharmacokinetics, biomarkers, and efficacy. No formal interim analyses will be performed.

Prior to enrollment, subjects will undergo screening to determine study eligibility. Upon enrollment, subjects will receive OMP-54F28 until disease progression. All subjects will receive Vitamin D3 daily and calcium carbonate twice daily from Day 0 through 30 days following the discontinuation of OMP-54F28.

Dose escalation will be conducted to determine the maximum tolerated dose (MTD). Subjects will be dosed at 0.5, 1, 2.5, 5, and 10 mg/kg administered IV once every 3 weeks. No dose escalation or reduction will be allowed within a dose cohort. Intermediate doses (i.e., doses between the dose levels listed above) may also be tested upon agreement with the investigators and the study sponsor. In addition, alternate dosing schedule cohorts of OMP-54F28 (eg. every 4 week or every 6 week dosing) can be studied upon agreement with the investigators and the study sponsor. These alternative less frequent dosing schedules may be evaluated if emerging data suggest that once every 3 week dosing results in tolerability concerns. The first 2 subjects enrolled in a cohort will not be treated on the same day. The dose may be administered at any time during the day. Three subjects will be treated at each dose level if no dose-limiting toxicities (DLTs) are observed. If 1 of 3 subjects experiences a DLT, that dose level will be expanded to 6 subjects. If 2 or more subjects experience a DLT, no further subjects will be dosed at that level and 3 additional subjects will be added to the preceding dose cohort unless 6 subjects have already been treated at that dose level. Subjects will be assessed for DLTs from Days 0-28. Dose escalation for newly enrolled subjects, if appropriate, will occur after all subjects in a cohort have completed their Day 28 DLT assessment. Subjects who have a >2-fold increase of their fasting β-CTX or a decline of >3% in their bone mineral density (BMD) from screening or a T-score decline to <-2.5 in the total femur or L1-L4 DEXA scan measurement will be started on zoledronic acid. Subjects with stable disease or a response at Day 56 will be allowed to continue to receive OMP-54F28 until disease progression. An additional 6 subjects will be enrolled in an expansion cohort at the highest dose level that results in <2 of the 6 subjects experiencing a Grade 3 (not including a Grade 3 infusion reaction that resolves in 24 hours) or Grade 4 adverse event (DLT). Tumors of particular interest for inclusion in the expansion cohort include sarcomas, basal cell carcinoma, ovarian cancer, desmoid tumors and prostate cancer given the known importance of the Wnt pathway in these malignancies.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be eligible for the study:

1. Subjects must have a histologically confirmed malignancy that is metastatic or unresectable and must have received the standard therapies for their malignancy. In addition, subjects must have a tumor that is at least 1 cm in a single dimension and is radiographically apparent on CT or MRI.
2. Subjects must have received their last chemotherapy, biologic, or investigational therapy at least 4 weeks prior to enrollment, 6 weeks if the last regimen included BCNU or mitomycin C.
3. Age >18 years
4. ECOG performance status <2 (see APPENDIX B)
5. Estimated life expectancy of more than 3 months
6. Subjects must have adequate organ and marrow function as defined below:

   Absolute neutrophil count >1000/µL Hemoglobin >9.0 g/dL Platelets >100,000/µL Total bilirubin <1.5 X institutional upper limit of normal (ULN) AST (SGOT) and ALT (SGPT) <3 X institutional ULN (for subjects with hepatic metastases <5 X institutional ULN) PT and PTT within 1.5 X institutional ULN Creatinine <1.5 X institutional ULN OR Creatinine clearance >60 mL/min/1.73 m2
7. Women of childbearing potential must have had a prior hysterectomy or have a negative serum pregnancy test and be using adequate contraception prior to study entry and must agree to use adequate contraception from study entry through at least 6 months after discontinuation of study drug. Men must also agree to use adequate contraception (barrier method of birth control, abstinence) prior to study entry and from study entry through at least 6 months after discontinuation of study drug. Should a woman enrolled in the study or a female partner of a man enrolled in the study become pregnant or suspect she is pregnant while participating in this study or within 6 months after discontinuation of study, she should inform the Investigator immediately.
8. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

Subjects who meet any of the following criteria will not be eligible for participation in the study:

1. Subjects receiving any other investigational agents
2. Subjects with brain metastases (subjects must have a CT scan or MRI of the head within 28 days prior to enrollment to rule out brain metastases), uncontrolled seizure disorder, or active neurologic disease
3. History of a significant allergic reaction attributed to humanized or human monoclonal antibody therapy or Fc fusion protein
4. Significant intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
5. Pregnant women or nursing women
6. Subjects with known HIV, Hepatitis B or Hepatitis C infection
7. Known bleeding disorder or coagulopathy
8. Subjects receiving heparin, warfarin, or other similar anticoagulants, except for subjects on low molecular weight heparin for DVT/PE prophylaxis. Note: Subjects may be receiving low-dose aspirin and/or non-steroidal anti-inflammatory agents.
9. New York Heart Association Classification III, or IV (see APPENDIX D)
10. Subjects with known clinically significant gastrointestinal disease including, but not limited to, inflammatory bowel disease.
11. Subjects with osteopenia or osteoporosis on their screening DEXA bone density scan.
12. Subjects with bone metastases that:

    1. have a prior history of a pathologic fracture,
    2. have a lytic lesion requiring an orthopedic intervention or
    3. are not receiving a bisphosphonate zoledronic acid or denosumab as per institutional guidelines All other subjects with bone metastases are eligible.
13. Subjects receiving a thiazolidinedione PPAR gamma inhibitor; i.e. Actos® (pioglitazone), Avandia® (rosiglitazone), and Rezulin® (troglitazone).
14. Subjects who have received ≥4 weeks of an oral or intravenous glucocorticoid at a dose that is equivalent to or greater than 5 mg of oral prednisone within the last 8 weeks.
15. Subjects with a fasting β-CTX of >1000 pg/mL.
16. Subjects with metabolic bone disease, such as hyperparathyroidism, Paget's disease or osteomalacia.
17. Subjects with a history of or a newly diagnosed insufficiency fracture or morphometric (asymptomatic) vertebral fracture on the screening lateral lumbosacral spine film.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-06; Primary Completion 2016-08 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
• To determine the safety of OMP-54F28 in subjects with previously treated solid tumors | Subjects will be assessed for dose limiting toxicities from Days 0-28. Adverse events will be reported through 30 days after the last dose.

SECONDARY OUTCOMES:
To determine the pharmacokinetics of OMP-54F28 in subjects with previously treated solid tumors | Baseline,end of infusion,0.5,1,3,6,24, and 72 hours post-infusion (1st infusion) 0.5, 1, 3, 6, 24, 72, and 168 hours (3rd infusion),before/end 2nd infusion,Days 7, 14, 28, and 35. After termination: Weekly for the first 4 weeks, then at Week 8 and 12
  The pharmacokinetic (PK) parameters to be assessed are study drug half-life (t½), volume of distribution (Vd), and clearance (CL).
To determine the immunogenicity of OMP-54F28 in subjects with previously treated solid tumors | Subjects will be assessed during screening ,every 4 weeks while on study drug, at the time of treatment termination, then weekly for the first 4 weeks, then at Week 8 and 12 following discontinuation of study drug
To assess the preliminary efficacy of OMP-54F28 in subjects with previously treated solid tumors | Every 56 days until disease progression
  The response outcome in patients will be determined.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Pinnacle Oncology Hematology,, Scottsdale, Arizona
  - University of Colorado Hospital, Aurora, Colorado
  - University of Michigan Health System, Ann Arbor, Michigan